CLINICAL TRIAL: NCT00098384
Title: A Randomized, Double-Blind, Single Center, Comparative Dose Ranging Study of Rifaximin Vs. Placebo in the Prevention of Travelers' Diarrhea Due to Enteropathogenic Bacteria
Brief Title: Rifaximin Versus Placebo in the Prevention of Travelers' Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DuPont, Hurbert L., MD (Individual)
Collaborators: Bausch Health Americas, Inc. (Industry); The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR 03
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2004-12

CONDITIONS: Diarrhea
Keywords: Travelers' diarrhea; rifaximin; prophylaxis; enterotoxigenic E. coli
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin

INTERVENTIONS:
Drug: rifaximin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of poorly absorbed rifaximin in the prevention of travelers' diarrhea among U.S. college students in Mexico for five weeks.

DETAILED DESCRIPTION:
This is an investigator-initiated proposal wherein 220 male and female subjects >17 years of age from industrialized regions were randomized to receive a poorly absorbed antibiotic, rifaximin, in one of three doses at mealtime (when they are exposed to diarrhea-causing bacteria), 200 mg once a day, 200 mg twice a day or 200 mg three times a day versus a placebo starting on arrival (within the first 72 hours) to Mexico and continuing for two weeks with diaries of symptoms recorded for three weeks. Adverse events in the subjects were followed for five weeks. If mild diarrhea (1 or 2 unformed stools/24 hours plus an enteric symptom) or diarrheal illness (>2 unformed stools/24 hours plus an enteric symptom) developed, subjects provided a stool sample to determine cause of illness. Forty subjects provided stool samples after 7 days and 14 days treatment to see if their intestinal bacterial flora had developed resistance to rifaximin and to see the level of drug achieved. Stool samples from these forty subjects were studied for enteric pathogens to look for asymptomatic infection during the period of prophylaxis. The stool samples collected were initially processed in our enteric laboratories in Guadalajara, Mexico. Specialized tests such as studies of toxigenicity for enterotoxigenic E. coli and enteroadherence for enteroaggregative E. coli were done in Houston.

ELIGIBILITY:
Inclusion Criteria:

* An Investigational Review Board approved, written informed consent is appropriately witnessed, signed and dated prior to any study-related activities
* Male or female subjects 18 years of age or older
* Able to read and understand English
* Enrolled and started on prophylaxis within 72 hours of arrival in Mexico
* If the subject is female, only women with non-childbearing potential or those who are not pregnant will be eligible. Urine pregnancy tests will be performed on those women who question their pregnancy status. Women on the study are required to employ a reliable method of contraception while taking medication. Forms of acceptable contraception include:

  * Double barrier method of contraception.
  * Oral birth control pills for at least two cycles before enrollment and continuing during therapy - subjects will be told they should use a barrier contraception method during the study as well.
  * Norplant inserted at least one month before enrollment.
  * An intrauterine device inserted by a qualified clinician.
  * Medroxyprogesterone acetate for a minimum of one month before study and administered for one month following study completion.
  * An approved birth control patch for at least two cycles before enrollment and continuing during therapy. OR
  * Complete abstinence from intercourse for the two weeks of medication.

Exclusion Criteria:

* Acute diarrhea (criteria for travelers' diarrhea above) within the past week
* Diarrhea developing within 24 hours of study enrollment
* In Mexico for more than 72 hours
* Receipt of one of the following classes of drugs: fluoroquinolone (any drug in class), macrolide or azalide or trimethoprim-sulfamethoxazole within the past week or during the three week study
* Receipt of other medication to decrease the occurrence of diarrhea (e.g. bismuth subsalicylate or lactobacillus preparations)
* For females, pregnancy or breast feeding during the three week study
* Receipt of antidiarrheal medication (loperamide, bismuth subsalicylate, kaopectate) within 24 hours of enrollment
* Hypersensitivity to rifaximin
* Unstable medical condition including chronic renal failure and insulin dependent diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2003-06; Study Completion 2003-09

PRIMARY OUTCOMES:
Occurrence of diarrhea, defined as passage of >2 unformed stools/24 hr plus one or more signs or symptoms of enteric infection

SECONDARY OUTCOMES:
Occurrence of mild diarrhea (1 or 2 unformed stools/24 hr plus a sign or symptom)
Treatment failure (not well in five days)
Occurrence of moderate to severe abdominal pain/cramps or intestinal gas related symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autonoma de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] DuPont HL, Jiang ZD, Ericsson CD, Adachi JA, Mathewson JJ, DuPont MW, Palazzini E, Riopel LM, Ashley D, Martinez-Sandoval F. Rifaximin versus ciprofloxacin for the treatment of traveler's diarrhea: a randomized, double-blind clinical trial. Clin Infect Dis. 2001 Dec 1;33(11):1807-15. doi: 10.1086/323814. Epub 2001 Oct 23. PMID 11692292
- [Background] DuPont HL, Ericsson CD. Prevention and treatment of traveler's diarrhea. N Engl J Med. 1993 Jun 24;328(25):1821-7. doi: 10.1056/NEJM199306243282507. No abstract available. PMID 8502272
- [Result] DuPont HL, Jiang ZD, Okhuysen PC, Ericsson CD, de la Cabada FJ, Ke S, DuPont MW, Martinez-Sandoval F. A randomized, double-blind, placebo-controlled trial of rifaximin to prevent travelers' diarrhea. Ann Intern Med. 2005 May 17;142(10):805-12. doi: 10.7326/0003-4819-142-10-200505170-00005. PMID 15897530